CLINICAL TRIAL: NCT02827084
Title: Effects of Kinesio Taping in Painful and Neuromuscular Performance of Patients With Patellofemoral Pain
Brief Title: Effects of Kinesio Taping in Patellofemoral Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20151012
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: electromyography; torque; quadriceps muscle
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kinesio Taping (Experimental): Apply the Kinesio Taping with tension in the vatus mediallis
  Interventions: Device: Kinesio Taping
- Placebo (Placebo Comparator): Apply the Kinesio Taping without tension in the vatus mediallis
  Interventions: Device: Placebo
- Control (No Intervention): It will not apply Kinesio.

INTERVENTIONS:
Device: Kinesio Taping — Application of the Kinesio Taping with tension in the vatus mediallis muscle.
  Other Names: Functional elastic tape
  Arms: Kinesio Taping
Device: Placebo — Application of the Kinesio Taping without tension in the vatus mediallis muscle.
  Other Names: Placebo functional elastic tape
  Arms: Placebo

SUMMARY:
The study aims to analyze the immediate effects and 72 hours after application of the Kinesio Taping (KT) in the electromyographic activity of the vastus medialis oblique (VMO) and vastus lateralis (VL), the isokinetic performance of the quadriceps and referred pain of subjects with PFPS. The volunteers will be randomly assigned to one of the three groups and perform one of the protocols: control - remain at rest; KT - application of Kinesio Taping with tension in the VMO region; placebo - application of Kinesio Taping without tension, in the same region. All volunteers will be submitted to the evaluation of pain intensity, the electromyographic activity of the VMO and VL and dynamometric parameters in 3 times: before the application of KT, immediately after the application of KT and after 72h of application. Average effect estimates (differences between groups) for all variables will be calculated using the mixed model ANOVA with a significance level of 5% (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 35 years;
* BMI below 30;
* Clinical diagnosis- previous pain or retropatellar in at least two of the following functional activities: stay for a long time sitting, up or down stairs, run, kneel, crouch, jump;
* Onset of symptoms insidiously and nontraumatic;
* Pain intensity 3 or more on EVA;
* Presence of pain for at least 1 month;

Exclusion Criteria:

* Be performing currently physiotherapy;
* It present surgery, trauma or musculoskeletal system of the lower limb injury within 6 months;
* There have other pathologies associated with the knee joint;
* Does not run the tests properly;
* Does not attend all assessments.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Onset of Electromyographic | Change from baseline in electromyographic at one hour and three days
  Evaluation of onset electromyographic activity of Vastus Medialis Obliquus relative to Vastus Lateralis

CONTACTS AND LOCATIONS:
Overall Officials: Jamilson S Brasileiro, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil